CLINICAL TRIAL: NCT00977938
Title: A Prospective, Multi-center, Randomized, Double-blind Trial to Assess the Effectiveness and Safety of 12 Versus 30 Months of Dual Antiplatelet Therapy in Subjects Undergoing Percutaneous Coronary Intervention With Either Drug-eluting Stent or Bare Metal Stent Placement for the Treatment of Coronary Artery Lesions
Brief Title: The Dual Antiplatelet Therapy Study (DAPT Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: Abbott (Industry); Boston Scientific Corporation (Industry); Bristol-Myers Squibb (Industry); Sanofi-Synthelabo (Industry); Cordis US Corp. (Industry); Eli Lilly and Company (Industry); Daiichi Sankyo (Industry); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HCRIG080186
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Results first posted 2015-10-22 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease
Keywords: Acute Coronary Syndrome; Adverse event; Antiplatelet therapy; Sirolimus; Everolimus; Paclitaxel; Zotarolimus; Bare Metal Stent; Drug Eluting Stent; Clinical Events Committee; Dual antiplatelet therapy; Harvard Clinical Research Institute; Major Adverse Cardiac and Cerebral Event; Major Bleeding; Myocardial infarction; Myocardial ischemia; Percutaneous coronary intervention; Stent placement; Stent Thrombosis; Thienopyridine; Clopidogrel; Prasugrel
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia | interventions — Aspirin; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12m DAPT Study Arm (Placebo Comparator): This population consists of subjects enrolled in the study who are free from death, MI, stroke, repeat coronary revascularization, major bleeding, and ST 12 months after stent implantation and who are compliant with 12 months of dual antiplatelet therapy following stent implantation and who are subsequently randomized to receive 18 months of placebo treatment in addition to aspirin.
  Interventions: Drug: Placebo & Aspirin
- 30m DAPT Study Arm (Active Comparator): This population consists of subjects enrolled in the study who are free from death, MI, stroke, repeat coronary revascularization, major bleeding, and ST 12 months after stent implantation and who are compliant with 12 months of dual antiplatelet therapy following stent implantation and who are subsequently randomized to receive an additional 18 months of thienopyridine treatment in addition to aspirin.
  Interventions: Drug: Clopidogrel & Aspirin, Prasugrel & Aspirin

INTERVENTIONS:
Drug: Placebo & Aspirin
  Arms: 12m DAPT Study Arm
Drug: Clopidogrel & Aspirin, Prasugrel & Aspirin
  Arms: 30m DAPT Study Arm

SUMMARY:
The DAPT Study is a double blind randomized controlled trial intended to determine the appropriate duration for dual antiplatelet therapy (the combination of aspirin and a second anti-clotting medication) as well as the safety and effectiveness of dual antiplatelet therapy to protect patients from stent thrombosis and major adverse cardiovascular and cerebrovascular events (MACCE) following the implantation of drug-eluting coronary stents. Similar analysis will be conducted in a smaller cohort of bare metal coronary stent - treated subjects.

DETAILED DESCRIPTION:
Subjects with ischemic heart disease due to stenotic lesions in either native coronary arteries or coronary artery bypass grafts undergoing percutaneous coronary intervention (PCI) with stent placement and no contraindications to prolonged dual antiplatelet therapy are eligible to be enrolled in the study.

All enrolled subjects will undergo PCI with stent placement. All enrolled subjects will be treated with either an FDA-approved drug eluting stent(s) (DES) or an FDA-approved bare metal stent(s) (BMS) (per their respective Instructions for Use) and assigned to 12 months of open label FDA-approved thienopyridine treatment in addition to aspirin. Operators will select the thienopyridine according to the package insert. Thienopyridine treatment dose will be according to the standard of practice and prescribing information for the selected medication. Aspirin treatment will be 75-325 mg for the first 6 months after the procedure and 75-162 mg subsequently, to be continued indefinitely. All DES or BMS subjects who are treated with 12 months of dual antiplatelet therapy post index procedure and who are event free per protocol will be eligible for randomization to either placebo (12 m DAPT Study arm) or an additional 18 months of thienopyridine treatment (30 m DAPT Study arm). Both arms will continue aspirin therapy.

Up to four (4) separate post-market approval studies will be allowed to incorporate the randomized design of the DAPT Study for a subset of subjects who may then be contributed for the DAPT Study analyses.

ELIGIBILITY:
Inclusion Criteria (Enrollment):

1. Subject is > 18 years of age.
2. Subjects undergoing percutaneous intervention with stent deployment (or has w/in 24 hours).
3. Subjects without known contraindication to dual antiplatelet therapy for at least 30 months after enrollment and stent implantation.
4. The subject has consented to participate and has authorized the collection and release of his medical information by signing the "Patient Informed Consent Form". The informed consent will be valid for the duration of the trial or until the subject withdraws.

Inclusion Criterion (Randomization at 12 months):

1. Subject, at 12 months, is free from death, MI, stroke, repeat coronary revascularization, major bleeding, and stent thrombosis and has been compliant with dual antiplatelet therapy following stent implantation.

Exclusion Criteria (Enrollment):

1. Index procedure stent placement with stent diameter <2.25 mm or >4.0 mm.
2. Pregnant women.
3. Planned surgery necessitating discontinuation of antiplatelet therapy within the 30 months following enrollment.
4. Current medical condition with a life expectancy of less than 3 years.
5. Concurrent enrollment in another device or drug study whose protocol specifically excludes concurrent enrollment or that involves blinded placement of a DES or BMS other than those included as DAPT Study devices. The subject may only be enrolled in the DAPT Study once.
6. Subjects on warfarin or similar anticoagulant therapy.
7. Subjects with hypersensitivity or allergies to one of the drugs or components indicated in the Instructions for Use for the device implanted.
8. Subjects unable to give informed consent.
9. Subject treated with both DES and BMS during the index procedure.

Exclusion Criteria (Randomization at 12 months):

1. Pregnant women.
2. Subject switched thienopyridine type or dose within 6 months prior to randomization.
3. Percutaneous coronary intervention or cardiac surgery between 6 weeks post index procedure and randomization.
4. Planned surgery necessitating discontinuation of antiplatelet therapy within the 21 months following randomization.
5. Current medical condition with a life expectancy of less than 3 years.
6. Subjects on warfarin or similar anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25682 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mauri, MD, MSc, Principal Investigator — Brigham and Women's Hospital; Dean Kereiakes, MD, FACC, Principal Investigator — Christ Hospital Heart and Vascular Center
Locations (255):
- United States (177):
  - Thomas Hospital, Fairhope, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Heart & Vascular Center of Arizona, Phoenix, Arizona
  - Scottsdale Health Care, Scottsdale, Arizona
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - University of Arkansas (Central VA) for Medical Science, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - California Cardiovascular Consultants/ Washington Hospital, Fremont, California
  - The Foundation for Cardiovascular Medicine, La Jolla, California
  - Mercy General Hospital, Sacramento, California
  - UC San Diego Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - St. Joseph's Medical Center- CA, Stockton, California
  - Torrance Memorial Medical Center / Vasek Polak Research Program, Torrance, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Medical Center of Aurora, Aurora, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - St. Vincent's Medical Center, Stamford, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Palm Beach Heart Research Institute, Atlantis, Florida
  - Bay Area Cardiology Associates/ Brandon Regional Hospital, Brandon, Florida
  - Jacksonville Heart Center, Jacksonville, Florida
  - Watson Clinic Center for Research, Lakeland, Florida
  - Diagnostic Cardiology Associates, Lauderdale Lakes, Florida
  - Melbourne Internal Medicine Assoc, Melbourne, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Munroe Regional Medical Center, Ocala, Florida
  - Ocala Regional Medical Center, Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Baptist Hospital, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Pepin Heart Hospital, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital Research Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Medical Center Central Georgia, Macon, Georgia
  - Redmond Regional Hospital, Rome, Georgia
  - Advocate Good Shephard Hospital, Barrington, Illinois
  - Jesse Brown VA Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Good Samaritan Hospital- IL, Downers Grove, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Heartland Education and Research Foundation, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Heart Care Research Foundation, Mokena, Illinois
  - Edward Heart Hospital, Naperville, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - St. Vincent Heart Center of Indiana, LLC, Indianapolis, Indiana
  - Northwest Indiana Cardiovascular Physicians, P.C., Valparaiso, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - St. Luke's Hospital - Cedar Rapids, Cedar Rapids, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - Kings Daughters Medical Center, Ashland, Kentucky
  - Tulane University Medical School, New Orleans, Louisiana
  - Northeast Cardiology Associates, Bangor, Maine
  - Maine Medical Center, Portland, Maine
  - Sinai Hospital at Baltimore, Baltimore, Maryland
  - Union Memorial Hospital, Baltimore, Maryland
  - Shah Associates, LLC, Prince Frederick, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Medical Center, Burlington, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Bay Regional Medical Center, Bay City, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital Heart & Vascular Institute, Detroit, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - St. Joseph Mercy-PTCMI, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Great Lakes Heart & Vascular Institute, PC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Beaumont Hospital Troy, Troy, Michigan
  - Mayo Clinic - Saint Marys Hospital, Rochester, Minnesota
  - Central Minnesota Heart Center at St. Cloud Hospital, Saint Cloud, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - St. Luke's Hospital Mid America Heart Institute, Kansas City, Missouri
  - Kansas City Heart Foundation, Kansas City, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - St. John's Medical Institute, Springfield, Missouri
  - Washington University Hospital, St Louis, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Alegent Health / Bergan Mercy Hospital, Omaha, Nebraska
  - Creighton University, Omaha, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Cardiovascular Associates of the Delaware Valley, PA, Haddon Heights, New Jersey
  - Hamilton Cardiology Associates, Hamilton, New Jersey
  - Valley Hospital, Hawthorne, New Jersey
  - UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Michaels Hospital, Newark, New Jersey
  - Presbyterian Heart Group, Albuquerque, New Mexico
  - SJH Cardiology Associates, Liverpool, New York
  - Winthrop University Hospital, Mineola, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - St. Elizabeth's Medical Center- NY, Utica, New York
  - Westchester Medical Center, Valhalla, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolina Heart Specialists, Gastonia, North Carolina
  - Carolina Cardiology Associates, High Point, North Carolina
  - Wake Heart Association, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - MeritCare Medical Center, Fargo, North Dakota
  - Altru Health System, Grand Forks, North Dakota
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Riverside Methodist, Columbus, Ohio
  - Elyria Memorial Hospital, Elyria, Ohio
  - Frederick C Smith Clinic dba Smith Clinic, Marion, Ohio
  - Northwest Ohio Cardiology, Toledo, Ohio
  - Midwest Regional Medical Center, Midwest City, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Foundation for CV Research, Oklahoma City, Oklahoma
  - St. Vincent Hospital/ Providence Heart Hospital, Portland, Oregon
  - Oregon Health & Sciences University Hospital, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Clinic, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pinnacle Health Hospital, Harrisburg, Pennsylvania
  - Conemaugh Memorial Medical Center, Johnstown, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Berks Cardiologists, Wyomissing, Pennsylvania
  - York Hospital (PA), York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Black Hills Research- Rapid City Regional, Rapid City, South Dakota
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Chattanooga Heart - East Third Street, Chattanooga, Tennessee
  - Chattanooga Heart Institute, Chattanooga, Tennessee
  - Centennial Heart Medical Center, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Capital Cardiovascular Research Institute, Austin, Texas
  - Texas Cardiovascular, Austin, Texas
  - Veteran's Affairs Medical Center- Dallas, Dallas, Texas
  - CRSTI Research, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - North Dallas Research Associates, McKinney, Texas
  - North Dallas Research Associate, McKinney, Texas
  - The Heart Hospital / Baylor Plano, Plano, Texas
  - Scott and White Healthcare - Round Rock, Round Rock, Texas
  - TexSan Heart Hospital, San Antonio, Texas
  - Mother Frances Hospital, Tyler, Texas
  - Providence Healthcare Network, Waco, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Rockingham Memorial Hospital, Harrisonburg, Virginia
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Sentara, Norfolk General Hospital, Norfolk, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Cardiovascular Associates, Ltd., Virginia Beach, Virginia
  - Winchester Medical Center, Winchester, Virginia
  - Providence St. Peter Hospital, Olympia, Washington
  - University of Washington, Seattle, Washington
  - Inland Cardiology Associates, Spokane, Washington
  - Sacred Heart Medical Center, Spokane, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - CaRE Foundation, Inc., Wausau, Wisconsin
- Australia (9):
  - St. Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Prince of Wales Eastern Heart, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Prahran, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - The Mount Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Monash Heart, Clayton
  - St Vincents Hospital Melbourne, Fitzroy
- Czechia (5):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Krajska karlovarska nemocnice a.s., Karlovy Vary
  - Centrum pro choroby srdce a cev, Kroměříž
  - Mestska nemocnice Ostrava, Ostrava
  - Krajska nemocnice T. Bati a.s., Zlín
- France (7):
  - Centre Hospitalier Saint Louis, La Rochelle
  - Hospital Saint Philibert, Lomme
  - Nouvelles Cliniques Nantaises, Nantes
  - Clinique les Franciscaines, Nîmes
  - Hopital Bichat, Paris
  - Groupe Hospitalier Sud, Pessac
  - CH Chatiliez Tourcoing, Tourcoing
- Germany (11):
  - Universitaetsklinikum Schleswig-Holstein - PS, Lübeck, Schleswig-Holstein
  - Helios Klinikum Emil von Behring, Berlin, State of Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Vivantes-Klinikum Neukoelin, Berlin
  - Vivantes-Klinikum Neukoelln, Berlin
  - Vivantes-Humboldt Klinikum, Berlin
  - Elbe-Kliniken Stade-Buxtehude GmbH, Buxtehude
  - Universitaetsklinikum Dresden, Dresden
  - Asklepios Klinik St. Georg, Hamburg
  - Herzzentrum Leipzig GmbH, Leipzig
  - Elbe-Kliniken Stade-Buxtehude GmbH, Stade
- Hungary (5):
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Josa Andras Oktato Korhaz Nonprofit Kft, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Klinikai Kozpont, Szeged
  - Zala Megyei Korhaz, Zalaegerszeg
- New Zealand (9):
  - Mercy Angiography, Epsom, Auckland
  - North Shore Hospital, Auckland
  - Ascot Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Nelson Hospital, Nelson
  - Wellington Hospital, Wellington
  - Wakefield Hospital, Wellington
- Poland (7):
  - Uniwersyteck Szpital Klin. w Bialymstoku, Bialystok
  - Wielospecj. Szpital Miejski im.dr.E.Warminskiego-SPZOZ, Bydgoszcz
  - NZOZ Centrum Medyczne Beluga-Med, Krakow
  - Szpital Uniwersytecki w Krakowie, Krakow
  - SPSK nr 2 Pomorskiej Akademii Medycznej w Szczecinie, Szczecin
  - Polsko-Amerykanskie Kliniki Serca.American Heart of Poland S, Ustroń
  - Instytut Kardiologii im. Kardynala St. Wyszynskiego, Warsaw
- Romania (7):
  - Centrul Clinic de Urgenta de Boli Cardiovasculare al Armatei, Bucharest
  - Spitalul Clinic de Urgenta Bucuresti, Bucharest
  - Inst. Urgenta Boli Cardiovasculare Prof. Dr. C.C. Iliescu, Bucharest
  - Institutul de Urgenta pentru Boli Cardiovasculare Prof. Dr., Bucharest
  - Spitalul Clinic Universitar de Urgenta Bucuresti, Bucharest
  - Institutul Inimii Niculae Stancioiu Cluj-Napoca, Cluj-Napoca
  - Institutul de Boli Cardiovasculare si Transplant Targu Mures, Târgu Mureş
- United Kingdom (18):
  - Wycombe General Hospital, High Wycombe, Bucks
  - Papworth Hospital, Cambridge, Cambs
  - Torbay hospital, Torquay, Devon
  - Royal Bournemouth General Hospital, Bournemouth, Dorset
  - Basildon University Hospital, Basildon, Essex
  - Barnet Hospital, Barnet, Herts
  - James Cook Hospital, Middlesbrough, N York
  - Ninewells Hospital, Dundee, Scotland
  - Weston General Hospital, Weston-super-Mare, Somerset
  - Golden Jubilee National Hospital, Glasgow, Strath
  - St Peter's Hospital, Chertsey
  - University Hospital of Coventry and Warwickshire, Coventry
  - Ninewells Hospital, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - University Hospital of Leicester Glenfield Hospital, Leicester
  - The London Chest Hospital, London
  - Freeman Hospital, Newcastle
  - Derriford Hospital, Plymouth

REFERENCES:
- [Derived] Faridi KF, Strom JB, Kundi H, Butala NM, Curtis JP, Gao Q, Song Y, Zheng L, Tamez H, Shen C, Secemsky EA, Yeh RW. Association Between Claims-Defined Frailty and Outcomes Following 30 Versus 12 Months of Dual Antiplatelet Therapy After Percutaneous Coronary Intervention: Findings From the EXTEND-DAPT Study. J Am Heart Assoc. 2023 Jul 18;12(14):e029588. doi: 10.1161/JAHA.123.029588. Epub 2023 Jul 14. PMID 37449567
- [Derived] Berg DD, Yeh RW, Mauri L, Morrow DA, Kereiakes DJ, Cutlip DE, Gao Q, Jarolim P, Michelson AD, Frelinger AL 3rd, Cange AL, Sabatine MS, O'Donoghue ML. Biomarkers of platelet activation and cardiovascular risk in the DAPT trial. J Thromb Thrombolysis. 2021 Apr;51(3):675-681. doi: 10.1007/s11239-020-02221-5. PMID 32683645
- [Derived] Stefanescu Schmidt AC, Steg PG, Yeh RW, Kereiakes DJ, Tanguay JF, Hsieh WH, Massaro JM, Mauri L, Cutlip DE; DAPT Investigators. Interruption of Dual Antiplatelet Therapy Within Six Months After Coronary Stents (from the Dual Antiplatelet Therapy Study). Am J Cardiol. 2019 Dec 15;124(12):1813-1820. doi: 10.1016/j.amjcard.2019.09.006. Epub 2019 Sep 26. PMID 31653353
- [Derived] Berry NC, Kereiakes DJ, Yeh RW, Steg PG, Cutlip DE, Jacobs AK, Abbott JD, Hsieh WH, Massaro JM, Mauri L; DAPT Study Investigators. Benefit and Risk of Prolonged DAPT After Coronary Stenting in Women. Circ Cardiovasc Interv. 2018 Aug;11(8):e005308. doi: 10.1161/CIRCINTERVENTIONS.117.005308. PMID 30354781
- [Derived] Yeh RW, Kereiakes DJ, Steg PG, Cutlip DE, Croce KJ, Massaro JM, Mauri L; DAPT Study Investigators. Lesion Complexity and Outcomes of Extended Dual Antiplatelet Therapy After Percutaneous Coronary Intervention. J Am Coll Cardiol. 2017 Oct 31;70(18):2213-2223. doi: 10.1016/j.jacc.2017.09.011. PMID 29073947
- [Derived] Secemsky EA, Yeh RW, Kereiakes DJ, Cutlip DE, Cohen DJ, Steg PG, Cannon CP, Apruzzese PK, D'Agostino RB Sr, Massaro JM, Mauri L; Dual Antiplatelet Therapy (DAPT) Study Investigators. Mortality Following Cardiovascular and Bleeding Events Occurring Beyond 1 Year After Coronary Stenting: A Secondary Analysis of the Dual Antiplatelet Therapy (DAPT) Study. JAMA Cardiol. 2017 May 1;2(5):478-487. doi: 10.1001/jamacardio.2017.0063. PMID 28297015
- [Derived] Stefanescu Schmidt AC, Kereiakes DJ, Cutlip DE, Yeh RW, D'Agostino RB Sr, Massaro JM, Hsieh WH, Mauri L; DAPT Investigators. Myocardial Infarction Risk After Discontinuation of Thienopyridine Therapy in the Randomized DAPT Study (Dual Antiplatelet Therapy). Circulation. 2017 May 2;135(18):1720-1732. doi: 10.1161/CIRCULATIONAHA.116.024835. Epub 2017 Feb 22. PMID 28228427
- [Derived] Resor CD, Nathan A, Kereiakes DJ, Yeh RW, Massaro JM, Cutlip DE, Gabriel Steg P, Hsieh WH, Mauri L; Dual Antiplatelet Therapy Study Investigators. Impact of Optimal Medical Therapy in the Dual Antiplatelet Therapy Study. Circulation. 2016 Oct 4;134(14):989-998. doi: 10.1161/CIRCULATIONAHA.116.024531. Epub 2016 Aug 30. PMID 27576774
- [Derived] Kereiakes DJ, Yeh RW, Massaro JM, Cutlip DE, Steg PG, Wiviott SD, Mauri L; DAPT Study Investigators. DAPT Score Utility for Risk Prediction in Patients With or Without Previous Myocardial Infarction. J Am Coll Cardiol. 2016 May 31;67(21):2492-502. doi: 10.1016/j.jacc.2016.03.485. Epub 2016 Apr 1. PMID 27046159
- [Derived] Yeh RW, Secemsky EA, Kereiakes DJ, Normand SL, Gershlick AH, Cohen DJ, Spertus JA, Steg PG, Cutlip DE, Rinaldi MJ, Camenzind E, Wijns W, Apruzzese PK, Song Y, Massaro JM, Mauri L; DAPT Study Investigators. Development and Validation of a Prediction Rule for Benefit and Harm of Dual Antiplatelet Therapy Beyond 1 Year After Percutaneous Coronary Intervention. JAMA. 2016 Apr 26;315(16):1735-49. doi: 10.1001/jama.2016.3775. PMID 27022822
- [Derived] Meredith IT, Tanguay JF, Kereiakes DJ, Cutlip DE, Yeh RW, Garratt KN, Lee DP, Steg PG, Weaver WD, Holmes DR Jr, Brindis RG, Trebacz J, Massaro JM, Hsieh WH, Mauri L; DAPT Study Investigators. Diabetes Mellitus and Prevention of Late Myocardial Infarction After Coronary Stenting in the Randomized Dual Antiplatelet Therapy Study. Circulation. 2016 May 3;133(18):1772-82. doi: 10.1161/CIRCULATIONAHA.115.016783. Epub 2016 Mar 18. PMID 26994121
- [Derived] Hermiller JB, Krucoff MW, Kereiakes DJ, Windecker S, Steg PG, Yeh RW, Cohen DJ, Cutlip DE, Massaro JM, Hsieh WH, Mauri L; DAPT Study Investigators. Benefits and Risks of Extended Dual Antiplatelet Therapy After Everolimus-Eluting Stents. JACC Cardiovasc Interv. 2016 Jan 25;9(2):138-47. doi: 10.1016/j.jcin.2015.10.001. PMID 26793956
- [Derived] Mauri L, Elmariah S, Yeh RW, Cutlip DE, Steg PG, Windecker S, Wiviott SD, Cohen DJ, Massaro JM, D'Agostino RB Sr, Braunwald E, Kereiakes DJ; DAPT Study Investigators. Causes of late mortality with dual antiplatelet therapy after coronary stents. Eur Heart J. 2016 Jan 21;37(4):378-85. doi: 10.1093/eurheartj/ehv614. Epub 2015 Nov 18. PMID 26586780
- [Derived] Kereiakes DJ, Yeh RW, Massaro JM, Driscoll-Shempp P, Cutlip DE, Steg PG, Gershlick AH, Darius H, Meredith IT, Ormiston J, Tanguay JF, Windecker S, Garratt KN, Kandzari DE, Lee DP, Simon DI, Iancu AC, Trebacz J, Mauri L; DAPT Study Investigators. Stent Thrombosis in Drug-Eluting or Bare-Metal Stents in Patients Receiving Dual Antiplatelet Therapy. JACC Cardiovasc Interv. 2015 Oct;8(12):1552-62. doi: 10.1016/j.jcin.2015.05.026. PMID 26493248
- [Derived] Yeh RW, Kereiakes DJ, Steg PG, Windecker S, Rinaldi MJ, Gershlick AH, Cutlip DE, Cohen DJ, Tanguay JF, Jacobs A, Wiviott SD, Massaro JM, Iancu AC, Mauri L; DAPT Study Investigators. Benefits and Risks of Extended Duration Dual Antiplatelet Therapy After PCI in Patients With and Without Acute Myocardial Infarction. J Am Coll Cardiol. 2015 May 26;65(20):2211-21. doi: 10.1016/j.jacc.2015.03.003. Epub 2015 Mar 15. PMID 25787199
- [Derived] Kereiakes DJ, Yeh RW, Massaro JM, Driscoll-Shempp P, Cutlip DE, Steg PG, Gershlick AH, Darius H, Meredith IT, Ormiston J, Tanguay JF, Windecker S, Garratt KN, Kandzari DE, Lee DP, Simon DI, Iancu AC, Trebacz J, Mauri L; Dual Antiplatelet Therapy (DAPT) Study Investigators. Antiplatelet therapy duration following bare metal or drug-eluting coronary stents: the dual antiplatelet therapy randomized clinical trial. JAMA. 2015 Mar 17;313(11):1113-21. doi: 10.1001/jama.2015.1671. PMID 25781440
- [Derived] Yeh RW, Czarny MJ, Normand SL, Kereiakes DJ, Holmes DR Jr, Brindis RG, Weaver WD, Rumsfeld JS, Roe MT, Kim S, Driscoll-Shempp P, Mauri L. Evaluating the generalizability of a large streamlined cardiovascular trial: comparing hospitals and patients in the dual antiplatelet therapy study versus the National Cardiovascular Data Registry. Circ Cardiovasc Qual Outcomes. 2015 Jan;8(1):96-102. doi: 10.1161/CIRCOUTCOMES.114.001239. Epub 2014 Nov 16. PMID 25399847
- [Derived] Mauri L, Kereiakes DJ, Yeh RW, Driscoll-Shempp P, Cutlip DE, Steg PG, Normand SL, Braunwald E, Wiviott SD, Cohen DJ, Holmes DR Jr, Krucoff MW, Hermiller J, Dauerman HL, Simon DI, Kandzari DE, Garratt KN, Lee DP, Pow TK, Ver Lee P, Rinaldi MJ, Massaro JM; DAPT Study Investigators. Twelve or 30 months of dual antiplatelet therapy after drug-eluting stents. N Engl J Med. 2014 Dec 4;371(23):2155-66. doi: 10.1056/NEJMoa1409312. Epub 2014 Nov 16. PMID 25399658
- [Derived] Matteau A, Yeh RW, Kereiakes D, Orav EJ, Massaro J, Steg PG, Normand SL, Cutlip DE, Mauri L. Frequency of the use of low- versus high-dose aspirin in dual antiplatelet therapy after percutaneous coronary intervention (from the Dual Antiplatelet Therapy study). Am J Cardiol. 2014 Apr 1;113(7):1146-52. doi: 10.1016/j.amjcard.2013.10.015. Epub 2013 Nov 8. PMID 24332248
- [Derived] Mauri L, Kereiakes DJ, Normand SL, Wiviott SD, Cohen DJ, Holmes DR, Bangalore S, Cutlip DE, Pencina M, Massaro JM. Rationale and design of the dual antiplatelet therapy study, a prospective, multicenter, randomized, double-blind trial to assess the effectiveness and safety of 12 versus 30 months of dual antiplatelet therapy in subjects undergoing percutaneous coronary intervention with either drug-eluting stent or bare metal stent placement for the treatment of coronary artery lesions. Am Heart J. 2010 Dec;160(6):1035-41, 1041.e1. doi: 10.1016/j.ahj.2010.07.038. PMID 21146655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 08/13/2009 and 07/01/2011, a total of 25682 patients were enrolled into the DAPT Study either by HCRI (NCT00977938; 14491 pts) or from 1 of 4 PMS studies: Abbott Xience V US (NCT01106534; 2998 pts), Boston Scientific Liberté PAS (NCT00997503; 3904 pts), Cordis CYPRESS (NCT00954707; 2029 pts) and Medtronic EDUCATE (NCT01069003; 2260 pts).
Groups:
- DES 30-month DAPT; DES 12-month DAPT: Of the 22,866 DES enrolled pts, a total of 9,961 pts underwent randomization at 12 months (4,941 to 12m DAPT and 5,020 to 30m DAPT).
- BMS 30-month DAPT; BMS 12-month DAPT: Of the 2,816 BMS enrolled pts, a total of 1,687 pts underwent randomization at 12 months (845 to 12-month DAPT and 842 to 30-month DAPT).
Period: Treatment (12-30 mo. Post Procedure)
Arm/Group | DES 30-month DAPT | DES 12-month DAPT | BMS 30-month DAPT | BMS 12-month DAPT
Started | 5020 | 4941 | 842 | 845
Completed | 4783 | 4716 | 796 | 784
Not Completed | 237 | 225 | 46 | 61
Not completed — Withdrawal by Subject | 132 | 116 | 13 | 20
Not completed — Lost to Follow-up | 88 | 91 | 30 | 37
Not completed — Other | 17 | 18 | 3 | 4
Period: Observation (30-33 mo. Post Procedure)
Arm/Group | DES 30-month DAPT | DES 12-month DAPT | BMS 30-month DAPT | BMS 12-month DAPT
Started | 4783 | 4716 | 796 | 784
Completed | 4732 | 4658 | 784 | 781
Not Completed | 51 | 58 | 12 | 3
Not completed — Withdrawal by Subject | 9 | 12 | 2 | 0
Not completed — Lost to Follow-up | 34 | 42 | 10 | 3
Not completed — Other | 8 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DES 30-month DAPT: Patients who were treated with DES at the index procedure and were randomized at 12 months post procedure to receive a total of 30 months of DAPT
- DES 12-month DAPT: Patients who were treated with DES at the index procedure and were randomized at 12 months post procedure to receive a total of 12 months of DAPT
- BMS 30-month DAPT: Patients who were treated with BMS at the index procedure and were randomized at 12 months post procedure to receive a total of 30 months of DAPT
- BMS 12-month DAPT: Patients who were treated with BMS at the index procedure and were randomized at 12 months post procedure to receive a total of 12 months of DAPT
- Total: Total of all reporting groups
Arm/Group | DES 30-month DAPT | DES 12-month DAPT | BMS 30-month DAPT | BMS 12-month DAPT | Total
Number analyzed (Participants) | 5020 | 4941 | 842 | 845 | 11648
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.84 (10.18) | 61.60 (10.12) | 58.86 (10.54) | 59.18 (11.07) | 61.33 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1242 | 1284 | 215 | 184 | 2925
  Male | 3778 | 3657 | 627 | 661 | 8723
Race/Ethnicity, Customized [Number; unit: participants] — Race was self-reported
  participants
    American Indian or Alaska Native | 17 | 41 | 0 | 2 | 60
    Asian | 48 | 35 | 3 | 2 | 88
    Black or African American | 252 | 253 | 38 | 33 | 576
    Native Hawaiian or Other Pacific Islander | 13 | 9 | 1 | 1 | 24
    White | 4480 | 4428 | 768 | 774 | 10450
    Other | 108 | 106 | 20 | 23 | 257
Region of Enrollment [Number; unit: participants]
  North America | 4502 | 4416 | 509 | 519 | 9946
  Europe | 402 | 405 | 304 | 300 | 1411
  Australia | 47 | 55 | 14 | 12 | 128
  New Zealand | 69 | 65 | 15 | 14 | 163
weight [Mean (Standard Deviation); unit: kg] | 91.49 (19.74) | 91.52 (19.43) | 87.99 (18.40) | 88.54 (18.77) | 91.04 (19.48)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.54 (5.79) | 30.55 (5.77) | 29.49 (5.18) | 29.61 (5.55) | 30.40 (5.73)
Diabetes Mellitus [Number; unit: participants] | 1556 | 1481 | 181 | 173 | 3391
Hypertension [Number; unit: participants] | 3796 | 3649 | 534 | 543 | 8522
Current cigarette smoker or within past year [Number; unit: participants] — "Current cigarette smoker or within past year" was defined as follows:
  * HCRI DAPT: current cigarette smoker or within past year
  * Abbott Xience V: current tobacco user or former tobacco user within the past month
  * Boston Scientific Liberte PAS: smoking status of "current" from medical history
  * Cordis CYPRESS: smoking within 30 days
  * Medtronic EDUCATE: smoking/tobacco usage = "current" or "within last year"
  participants | 1222 | 1210 | 360 | 350 | 3142
Stroke/Transient Ischemic Attack (TIA) [Number; unit: participants] | 155 | 169 | 43 | 34 | 401
Congestive heart failure [Number; unit: participants] | 238 | 223 | 35 | 28 | 524
Peripheral arterial disease [Number; unit: participants] | 284 | 284 | 35 | 46 | 649
Prior percutaneous coronary intervention (PCI) [Number; unit: participants] | 1518 | 1529 | 150 | 171 | 3368
Prior coronary artery bypass graf (CABG) [Number; unit: participants] | 568 | 581 | 50 | 50 | 1249
Prior myocardial infarction (MI) [Number; unit: participants] | 1092 | 1026 | 160 | 178 | 2456
Indication for PCI [Number; unit: participants] — "Unstable angina" includes unstable angina without reported elevation of cardiac enzymes
  participants
    ST elevation MI (STEMI) | 534 | 511 | 311 | 324 | 1680
    Non-ST elevation MI (NSTEMI) | 776 | 767 | 184 | 169 | 1896
    Unstable angina | 838 | 825 | 77 | 81 | 1821
    Stable angina | 1882 | 1870 | 199 | 198 | 4149
    Other | 990 | 968 | 71 | 73 | 2102
Any risk factor for stent thrombosis [Number; unit: participants] — Any clinical or lesion-related risk factors for stent thrombosis.
  Clinical risk factors for stent thrombosis included:
  * Acute coronary syndrome (ACS) at presentation
  * ST elevation MI (STEMI) at presentation
  * Renal insufficiency or failure
  * Ejection fraction <30%.
  Lesion-related risk factors for stent thrombosis included:
  * More than two vessels stented
  * >2 lesions per vessel
  * Lesion length ≥30 mm
  * Bifurcation lesion with side branch ≥2.5 mm
  * In-stent restenosis of a DES
  * Vein bypass graft
  * Unprotected left main
  * Thrombus containing lesion
  * Prior brachytherapy
  participants | 2410 | 2389 | 568 | 569 | 5936
Number of treated lesions (per-patient) [Mean (Standard Deviation); unit: lesions] | 1.30 (0.55) | 1.29 (0.54) | 1.16 (0.40) | 1.17 (0.42) | 1.28 (0.53)
Number of treated vessels (per-patient) [Mean (Standard Deviation); unit: vessels] | 1.11 (0.33) | 1.12 (0.34) | 1.03 (0.18) | 1.05 (0.23) | 1.11 (0.32)
Number of stents (per-patient) [Mean (Standard Deviation); unit: stents] | 1.47 (0.75) | 1.45 (0.75) | 1.32 (0.60) | 1.32 (0.60) | 1.44 (0.73)
Minimum stent diameter (per-patient) [Number; unit: participants]
  <3 mm | 2341 | 2293 | 201 | 206 | 5041
  ≥3 mm | 2679 | 2648 | 641 | 639 | 6607
Total stent length (per-patient) [Mean (Standard Deviation); unit: mm] | 27.70 (16.77) | 27.43 (17.02) | 23.96 (13.01) | 23.85 (13.12) | 27.04 (16.44)
Treated Vessel [Number; unit: lesions] — The 5,020 DES 30-month DAPT patients had a total of 6,594 lesions; The 4,941 DES 12-month DAPT patients had a total of 6,413 lesions; The 842 BMS 30-month DAPT patients had a total of 975 lesions; The 845 BMS 12-month DAPT patients had a total of 991 lesions
  lesions
    Left main | 55 | 55 | 0 | 1 | 111
    Left anterior descending (LAD) | 2715 | 2586 | 308 | 306 | 5915
    Right coronary artery (RCA) | 2153 | 2057 | 437 | 452 | 5099
    Circumflex | 1473 | 1506 | 206 | 207 | 3392
    Venous graft | 154 | 173 | 24 | 25 | 376
    Arterial graft | 36 | 30 | 0 | 0 | 66
Modified ACC-AHA lesion class B2 or C [Number; unit: lesions] — The 5,020 DES 30-month DAPT patients had a total of 6,594 lesions; The 4,941 DES 12-month DAPT patients had a total of 6,413 lesions; The 842 BMS 30-month DAPT patients had a total of 975 lesions; The 845 BMS 12-month DAPT patients had a total of 991 lesions; The definitions of class B2 and class C lesions according to the modified ACC/AHA criteria
  lesions | 2754 | 2643 | 440 | 450 | 6287

OUTCOME MEASURES:

1. Primary Outcome: MACCE (Death, Myocardial Infarction or Stroke) - Randomized DES ITT
Description: The coprimary efficacy endpoints were the cumulative incidence of MACCE and the cumulative incidence of ARC definite or probable stent thrombosis within randomized DES ITT patients between 12 and 30 months post procedure.
Time Frame: 18 months (12-30 months post-index procedure)
Population: All randomized DES ITT patients; Patients were analyzed according to the treatment to which they were randomized (regardless of post-randomization compliance with the randomized treatment); Patients not experiencing the endpoint were censored at 30 months or at last known follow-up, whichever was earlier.
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | DES 30-month DAPT | DES 12-month DAPT
Number analyzed (Participants) | 5020 | 4941
percentage of patients (KM estimate) | 4.34 | 5.92
Statistical Analysis 1: Comparison: DES 30-month DAPT vs DES 12-month DAPT; The primary efficacy analysis was a superiority analysis. We controlled the two-sided family-wise error rate of 0.05 across the two coprimary end points using the Hochberg-Benjamini method. With this method, the null hypothesis of randomized treatment equivalence is rejected if significance is achieved for both end points at a two-sided alpha level of 0.05 or for one end point at a two-sided alpha level of 0.025; Test type: Superiority or Other; p < 0.001, Log Rank — P-value was stratified according to geographic region (NA, EU, or AU and NZ), thienopyridine received at the time of randomization, and presence or absence of risk factors for ST; P-value was adjudsted using the Benjamini Hochberg approach; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.59 to 0.85] — 30-month DAPT vs. 12-month DAPT; HR was stratified according to geographic region (NA, EU, or AU and NZ), thienopyridine drug received at the time of randomization, and presence or absence of risk factors for stent thrombosis

2. Primary Outcome: Definite or Probable Stent Thrombosis (ST) - Randomized DES ITT
Description: The coprimary efficacy endpoints were the cumulative incidence of MACCE and the cumulative incidence of definite or probable ST within randomized DES ITT patients between 12 and 30 months post procedure. ST was assessed according to the Academic Research Consortium (ARC) definitions.
Time Frame: 18 months (12-30 months post-index procedure)
Population: as for outcome 1
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | DES 30-month DAPT | DES 12-month DAPT
Number analyzed (Participants) | 5020 | 4941
percentage of patients (KM estimate) | 0.40 | 1.35
Statistical Analysis 1: Comparison: DES 30-month DAPT vs DES 12-month DAPT; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.17 to 0.48] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: GUSTO Severe or Moderate Bleeding - Randomized DES ITT
Description: The primary safety endpoint was moderate or severe bleeding within randomized DES ITT patients between 12 and 30 months post procedure. Bleeding was assessed according to the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Arteries (GUSTO) criteria.
Time Frame: 18 months (12-30 months post-index procedure)
Population: Only patients who could be evaluated were included in this analysis (i.e., patients whose last contact date was ≥510 days after randomization or who had any adjudicated bleeding event at or before 540 days).
Measure: Number; unit: percentage of patients
Arm/Group | DES 30-month DAPT | DES 12-month DAPT
Number analyzed (Participants) | 4710 | 4649
percentage of patients | 2.53 | 1.57
Statistical Analysis 1: Comparison: DES 30-month DAPT vs DES 12-month DAPT; Test type: Non-Inferiority or Equivalence — The primary safety analysis was a noninferiority analysis performed with the use of the Farrington-Manning risk-difference approach. Assuming an annualized rate for moderate or severe bleeding of 1.9% and an absolute noninferiority margin of 0.8%, at a one-sided alpha level of significance of 0.025, we calculated that a sample size of 9960 patients would give the study 80% power to detect noninferiority; p = 0.704, Farrington-Manning — One-sided P-value for non-inferiority; Risk Difference (RD) = 0.96, 95% CI 2-sided [0.38 to 1.53] — 30-month DAPT vs. 12-month DAPT

4. Secondary Outcome: MACCE (Death, Myocardial Infarction or Stroke) - Propensity Matched DES vs. BMS
Description: Secondary powered endpoint
Time Frame: 33 months (0-33 months post-index procedure)
Population: A subsample created by matching BMS- to DES-treated patients exactly on prevalence of STEMI and then matching on remaining baseline characteristics via propensity score, using a caliper width of 0.10. A BMS-treated patient was matched to a variable number of DES-treated patients without replacement, up to a maximum of 8.
Measure: Number; unit: percentage of patients
Groups:
- Propensity-matched DES: Because patients were not randomized to DES or BMS, DES comparisons vs. BMS on stent thrombosis and MACCE were carried out on sample matched on baseline characteristics via propensity score matching. The analyses were restricted to patients enrolled into the 3 contributing studies that planned to follow all enrolled patients (whether or not a patient was randomized) for 33 months. Patients prematurely withdrawing before 29 months follow-up (earliest allowable follow-up time for the 30-month visit) or before experiencing the endpoint were excluded. A total of 13,257 DES-treated patients were eligible for propensity matching, of whom 8,308 patients were matched to BMS-treated patients (up to 8 DES patients could be matched to a BMS patient; i.e., the BMS:DES matching ratio ranged from 1:1 to 1:8).
- Propensity-matched BMS: Because patients were not randomized to DES or BMS, DES comparisons vs. BMS on stent thrombosis and MACCE were carried out on sample matched on baseline characteristics via propensity score matching. The analyses were restricted to patients enrolled into the 3 contributing studies that planned to follow all enrolled patients (whether or not a patient was randomized) for 33 months. Patients prematurely withdrawing before 29 months follow-up (earliest allowable follow-up time for the 30-month visit) or before experiencing the endpoint were excluded. A total of 2,056 BMS-treated patients were eligible for propensity matching, of whom 1,718 were matched to at least one DES-treated patient (a BMS patient could be matched to up to 8 DES patients; i.e., the BMS:DES matching ratio ranged from 1:1 to 1:8).
Arm/Group | Propensity-matched DES | Propensity-matched BMS
Number analyzed (Participants) | 8308 | 1718
percentage of patients | 11.37 | 13.24
Statistical Analysis 1: Comparison: Propensity-matched DES vs Propensity-matched BMS; The null hypothesis was that DAPT patients treated with DES would have MACCE rate between 0 and 33 months post-index procedure that exceeds that of the control arm (patients treated with BMS) by at least a pre-specified absolute margin of δ; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 2.28% (0.0228); p < 0.001, Nam and Kwon — One-sided P-value for non-inferiority; P-value was computed for clustered matched pairs based on Nam and Kwon (2009); Risk Difference (RD) = -1.82, 97.5% CI 1-sided [upper limit 0.03] — Weighted RD and 1-sided 97.5% upper CL were computed for clustered matched pairs based on Nam and Kwon (2009)

5. Secondary Outcome: Definite or Probable Stent Thrombosis (ST) - Propensity Matched DES vs. BMS
Description: Secondary powered endpoint
Time Frame: 33 months (0-33 months post-index procedure)
Population: as for outcome 4
Measure: Number; unit: percentage of patients
Arm/Group | Propensity-matched DES | Propensity-matched BMS
Number analyzed (Participants) | 8308 | 1718
percentage of patients | 1.70 | 2.61
Statistical Analysis 1: Comparison: Propensity-matched DES vs Propensity-matched BMS; The null hypothesis was that DAPT patients treated with DES would have stent thrombosis rate between 0 and 33 months post-index procedure that exceeds that of the control arm (patients treated with BMS) by at least a pre-specified absolute margin of δ; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 0.97% (0.0097); p < 0.001, Nam and Kwon — One-sided P-value for non-inferiority; P-value was computed for clustered matched pairs based on Nam and Kwon (2009); Risk Difference (RD) = -1.05, 97.5% CI 1-sided [upper limit -0.27] — Weighted RD and 1-sided 95% upper CL were computed for clustered matched pairs based on Nam and Kwon (2009)

6. Secondary Outcome: MACCE (Death, Myocardial Infarction or Stroke) - Randomized DES ITT
Time Frame: 21 months (12-33 months post-index procedure)
Population: All randomized DES ITT patients; Patients were analyzed according to the treatment to which they were randomized (regardless of post-randomization compliance with the randomized treatment); Patients not experiencing the endpoint were censored at 33 months or at last known follow-up, whichever was earlier.
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | DES 30-month DAPT | DES 12-month DAPT
Number analyzed (Participants) | 5020 | 4941
percentage of patients (KM estimate) | 5.62 | 6.49
Statistical Analysis 1: Comparison: DES 30-month DAPT vs DES 12-month DAPT; Test type: Superiority or Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.70 to 0.97] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Definite or Probable Stent Thrombosis (ST) - Randomized DES ITT
Description: ST was assessed according to the Academic Research Consortium (ARC) definitions.
Time Frame: 21 months (12-33 months post-index procedure)
Population: as for outcome 6
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | DES 30-month DAPT | DES 12-month DAPT
Number analyzed (Participants) | 5020 | 4941
percentage of patients (KM estimate) | 0.69 | 1.45
Statistical Analysis 1: Comparison: DES 30-month DAPT vs DES 12-month DAPT; Test type: Superiority or Other; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.29 to 0.69] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: GUSTO Severe or Moderate Bleeding - Randomized DES ITT
Description: Bleeding was assessed according to the Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Arteries (GUSTO) criteria.
Time Frame: 21 months (12-33 months post-index procedure)
Population: Only patients who could be evaluated were included in this analysis (i.e., patients whose last contact date was ≥600 days after randomization or who had any adjudicated bleeding event at or before 630 days).
Measure: Number; unit: percentage of patients
Arm/Group | DES 30-month DAPT | DES 12-month DAPT
Number analyzed (Participants) | 4525 | 4476
percentage of patients | 2.74 | 1.88
Statistical Analysis 1: Comparison: DES 30-month DAPT vs DES 12-month DAPT; Test type: Superiority or Other; Risk Difference (RD) = 0.86, 95% CI 2-sided [0.24 to 1.48] — 30-month DAPT vs. 12-month DAPT

9. Secondary Outcome: MACCE (Death, Myocardial Infarction or Stroke) - Randomized BMS ITT
Time Frame: 18 months (12-30 months post-index procedure)
Population: All randomized BMS ITT patients; Patients were analyzed according to the treatment to which they were randomized (regardless of post-randomization compliance with the randomized treatment); Patients not experiencing the endpoint were censored at 30 months or at last known follow-up, whichever was earlier.
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | BMS 30-month DAPT | BMS 12-month DAPT
Number analyzed (Participants) | 842 | 845
percentage of patients (KM estimate) | 4.04 | 4.69
Statistical Analysis 1: Comparison: BMS 30-month DAPT vs BMS 12-month DAPT; This analysis was not powered; Test type: Superiority or Other; p = 0.722, Log Rank — This analysis was not powered. P-value was stratified according to geographic region, thienopyridine received at the time of randomization, and presence or absence of risk factors for ST; P-value was adjudsted using the Benjamini Hochberg approach; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.57 to 1.47] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Definite or Probable Stent Thrombosis (ST) - Randomized BMS ITT
Description: ST was assessed according to the Academic Research Consortium (ARC) definitions.
Time Frame: 18 months (12-30 months post-index procedure)
Population: as for outcome 9
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | BMS 30-month DAPT | BMS 12-month DAPT
Number analyzed (Participants) | 842 | 845
percentage of patients (KM estimate) | 0.50 | 1.11
Statistical Analysis 1: Comparison: BMS 30-month DAPT vs BMS 12-month DAPT; This analysis was not powered; Test type: Superiority or Other; p = 0.478, Log Rank — [p-value comment as in outcome 9, analysis 1]; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.15 to 1.64] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: GUSTO Severe or Moderate Bleeding - Randomized BMS ITT
Description: as for outcome 8
Time Frame: 18 months (12-30 months post-index procedure)
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | BMS 30-month DAPT | BMS 12-month DAPT
Number analyzed (Participants) | 790 | 776
percentage of patients | 2.03 | 0.90
Statistical Analysis 1: Comparison: BMS 30-month DAPT vs BMS 12-month DAPT; Test type: Superiority or Other; p = 0.706, Farrington-Manning; No formal hypothesis testing was done; Risk Difference (RD) = 1.12, 95% CI 2-sided [-0.06 to 2.31] — 30-month DAPT vs. 12-month DAPT

12. Secondary Outcome: MACCE (Death, Myocardial Infarction or Stroke) - Randomized BMS ITT
Time Frame: 21 months (12-33 months post-index procedure)
Population: All randomized BMS ITT patients; Patients were analyzed according to the treatment to which they were randomized (regardless of post-randomization compliance with the randomized treatment); Patients not experiencing the endpoint were censored at 33 months or at last known follow-up, whichever was earlier.
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | BMS 30-month DAPT | BMS 12-month DAPT
Number analyzed (Participants) | 842 | 845
percentage of patients (KM estimate) | 4.68 | 5.48
Statistical Analysis 1: Comparison: BMS 30-month DAPT vs BMS 12-month DAPT; Test type: Superiority or Other; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.58 to 1.40] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Definite or Probable Stent Thrombosis (ST) - Randomized BMS ITT
Description: ST was assessed according to the Academic Research Consortium (ARC) definitions.
Time Frame: 21 months (12-33 months post-index procedure)
Population: as for outcome 12
Measure: Number; unit: percentage of patients (KM estimate)
Arm/Group | BMS 30-month DAPT | BMS 12-month DAPT
Number analyzed (Participants) | 842 | 845
percentage of patients (KM estimate) | 0.50 | 1.11
Statistical Analysis 1: Comparison: BMS 30-month DAPT vs BMS 12-month DAPT; Test type: Superiority or Other; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.15 to 1.64] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: GUSTO Severe or Moderate Bleeding - Randomized BMS ITT
Description: as for outcome 8
Time Frame: 21 months (12-33 months post-index procedure)
Population: as for outcome 8
Measure: Number; unit: percentage of patients
Arm/Group | BMS 30-month DAPT | BMS 12-month DAPT
Number analyzed (Participants) | 766 | 759
percentage of patients | 2.09 | 1.05
Statistical Analysis 1: Comparison: BMS 30-month DAPT vs BMS 12-month DAPT; Test type: Superiority or Other; Risk Difference (RD) = 1.03, 95% CI 2-sided [-0.21 to 2.28] — 30-month DAPT vs. 12-month DAPT

ADVERSE EVENTS:
Time Frame: 12-33 months post-index procedure (randomization to 33 months post-index procedure)
Groups:
- HCRI DAPT - DES 30-month DAPT: Patients who were enrolled by HCRI into the HCRI DAPT Study, treated with DES at the index procedure and randomized at 12 months post procedure to receive a total of 30 months of DAPT
- HCRI DAPT - DES 12-month DAPT: Patients who were enrolled by HCRI into the HCRI DAPT Study, treated with DES at the index procedure and randomized at 12 months post procedure to receive a total of 12 months of DAPT
- HCRI DAPT - BMS 30-month DAPT: Patients who were enrolled by HCRI into the HCRI DAPT Study, treated with BMS at the index procedure and randomized at 12 months post procedure to receive a total of 30 months of DAPT
- HCRI DAPT - BMS 12-month DAPT: Patients who were enrolled by HCRI into the HCRI DAPT Study, treated with BMS at the index procedure and randomized at 12 months post procedure to receive a total of 12 months of DAPT
Arm/Group | HCRI DAPT - DES 30-month DAPT | HCRI DAPT - DES 12-month DAPT | HCRI DAPT - BMS 30-month DAPT | HCRI DAPT - BMS 12-month DAPT
Serious Adverse Events (participants affected / at risk) | 617/2642 | 572/2634 | 144/842 | 150/845
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCRI DAPT - DES 30-month DAPT (N=2642) | HCRI DAPT - DES 12-month DAPT (N=2634) | HCRI DAPT - BMS 30-month DAPT (N=842) | HCRI DAPT - BMS 12-month DAPT (N=845)
ANAEMIA (Blood and lymphatic system disorders) | 12 | 9 | 1 | 1
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
COAGULOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 3 | 1 | 0
RETROPERITONEAL LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 55 | 55 | 13 | 18
ANGINA UNSTABLE (Cardiac disorders) | 27 | 40 | 4 | 5
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 3 | 0 | 0 | 0
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 1 | 0 | 0 | 1
ARTERIOSPASM CORONARY (Cardiac disorders) | 0 | 1 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 24 | 14 | 3 | 9
ATRIAL FLUTTER (Cardiac disorders) | 2 | 6 | 1 | 0
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 1 | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0 | 0 | 0
BRADYCARDIA (Cardiac disorders) | 2 | 5 | 1 | 2
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 0 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 8 | 9 | 2 | 0
CARDIAC DISORDER (Cardiac disorders) | 0 | 0 | 1 | 1
CARDIAC FAILURE (Cardiac disorders) | 5 | 7 | 2 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1 | 2 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 22 | 14 | 4 | 5
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 2 | 1 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 22 | 16 | 9 | 6
CORONARY ARTERY DISSECTION (Cardiac disorders) | 0 | 1 | 0 | 0
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2 | 1 | 1 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 5 | 7 | 0 | 1
EXTRASYSTOLES (Cardiac disorders) | 1 | 0 | 0 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 2 | 0 | 1 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 1 | 0 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 0 | 0
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 1 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 1 | 0 | 5
PALPITATIONS (Cardiac disorders) | 1 | 4 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0 | 0
PERICARDITIS (Cardiac disorders) | 1 | 1 | 1 | 0
SICK SINUS SYNDROME (Cardiac disorders) | 2 | 0 | 2 | 1
SUBENDOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 0 | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 4 | 2 | 0 | 2
TACHYCARDIA (Cardiac disorders) | 1 | 1 | 0 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 | 2 | 0 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 4 | 0 | 1
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
HYDROCELE (Congenital, familial and genetic disorders) | 1 | 1 | 0 | 0
MYOTONIC DYSTROPHY (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
EXOSTOSIS OF EXTERNAL EAR CANAL (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
MENIERE'S DISEASE (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 2 | 5 | 0 | 0
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 1 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0 | 0 | 0
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 | 1 | 0 | 0
THYROID MASS (Endocrine disorders) | 0 | 1 | 0 | 0
CATARACT (Eye disorders) | 2 | 0 | 1 | 0
EYE PAIN (Eye disorders) | 0 | 1 | 0 | 0
GLAUCOMA (Eye disorders) | 0 | 0 | 0 | 1
MACULAR DEGENERATION (Eye disorders) | 0 | 1 | 0 | 0
RETINAL DETACHMENT (Eye disorders) | 0 | 1 | 1 | 0
RETINAL HAEMORRHAGE (Eye disorders) | 0 | 0 | 0 | 1
VISUAL ACUITY REDUCED (Eye disorders) | 2 | 0 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 1 | 1 | 3
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 1 | 2 | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 2 | 1 | 1 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 2 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 1 | 2 | 1
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DIVERTICULUM (Gastrointestinal disorders) | 0 | 1 | 0 | 0
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DUODENITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
EPIPLOIC APPENDAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 2 | 0 | 1 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 10 | 2 | 0 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 2 | 3 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 2 | 0 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 3 | 3 | 2 | 2
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 1 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 0 | 2
OESOPHAGEAL PERFORATION (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 1
PANCREATIC MASS (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PANCREATIC PSEUDOCYST (Gastrointestinal disorders) | 0 | 1 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 2 | 2 | 1 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 3 | 3 | 0 | 1
PHARYNGOESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1 | 0 | 0 | 0
POLYP COLORECTAL (Gastrointestinal disorders) | 0 | 1 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 1 | 0
RECTAL POLYP (Gastrointestinal disorders) | 1 | 1 | 0 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 5 | 1 | 0
SPIGELIAN HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 2 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0
VOLVULUS (Gastrointestinal disorders) | 0 | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 1
ADVERSE DRUG REACTION (General disorders) | 0 | 1 | 0 | 0
ASTHENIA (General disorders) | 1 | 1 | 0 | 0
CHEST DISCOMFORT (General disorders) | 8 | 4 | 0 | 1
CHEST PAIN (General disorders) | 43 | 45 | 12 | 7
DEATH (General disorders) | 1 | 1 | 0 | 0
HERNIA (General disorders) | 1 | 0 | 2 | 0
HERNIA OBSTRUCTIVE (General disorders) | 0 | 2 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 54 | 51 | 12 | 15
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 0 | 0
PAIN (General disorders) | 4 | 1 | 0 | 0
PELVIC MASS (General disorders) | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 1 | 1 | 0
SWELLING (General disorders) | 3 | 0 | 0 | 0
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 | 0 | 0 | 0
ALCOHOLIC LIVER DISEASE (Hepatobiliary disorders) | 1 | 0 | 0 | 1
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 1 | 0 | 0 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 1 | 0 | 0
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 0 | 0 | 1
BILIARY COLIC (Hepatobiliary disorders) | 0 | 2 | 0 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 5 | 2 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 7 | 7 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 2 | 3 | 0 | 1
CHOLESTASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHRONIC HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
ALLERGY TO METALS (Immune system disorders) | 0 | 0 | 0 | 1
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
ABSCESS (Infections and infestations) | 0 | 2 | 0 | 1
ABSCESS LIMB (Infections and infestations) | 1 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 7 | 1 | 0 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 1 | 1 | 0 | 0
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 2 | 1 | 1 | 0
BRONCHIECTASIS (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 5 | 5 | 2 | 0
BRONCHITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 2 | 0 | 0 | 0
CAMPYLOBACTER INTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 8 | 9 | 1 | 2
CELLULITIS STAPHYLOCOCCAL (Infections and infestations) | 0 | 1 | 0 | 0
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 | 1 | 0 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 0 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 6 | 6 | 1 | 3
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
GALLBLADDER ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0
GANGRENE (Infections and infestations) | 2 | 0 | 0 | 0
GASTRIC INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 3 | 2 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 2 | 1 | 0 | 0
GIARDIASIS (Infections and infestations) | 1 | 0 | 0 | 0
INFECTION (Infections and infestations) | 2 | 1 | 0 | 0
INFLUENZA (Infections and infestations) | 2 | 0 | 0 | 0
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1 | 0 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 2 | 2 | 0 | 0
MASTOIDITIS (Infections and infestations) | 1 | 0 | 0 | 0
MENINGITIS ASEPTIC (Infections and infestations) | 1 | 0 | 0 | 1
NEUTROPENIC SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
OSTEOMYELITIS (Infections and infestations) | 2 | 2 | 0 | 0
PANCREATIC ABSCESS (Infections and infestations) | 0 | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0
PILONIDAL CYST (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 21 | 17 | 4 | 4
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 0 | 0 | 0
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0
PSEUDOMONAS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 3 | 0 | 0 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 9 | 7 | 1 | 0
SEPSIS SYNDROME (Infections and infestations) | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 0 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
STITCH ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 5 | 7 | 2 | 1
UROSEPSIS (Infections and infestations) | 3 | 0 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 3 | 0 | 0
WOUND INFECTION (Infections and infestations) | 1 | 1 | 0 | 0
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
COLLAPSE OF LUNG (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
CONTUSION (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
DEVICE MALFUNCTION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 4 | 2 | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
IN-STENT ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 1
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 11 | 5 | 4 | 2
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
INJURY (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
MENISCUS LESION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
PUBIC RAMI FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
TENDON INJURY (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
THROMBOSIS IN DEVICE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
URETHRAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
URINARY BLADDER RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
VASCULAR BYPASS DYSFUNCTION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
VASCULAR GRAFT OCCLUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
ANTIMICROBIAL SUSCEPTIBILITY TEST RESISTANT (Investigations) | 0 | 1 | 0 | 0
BLOOD CREATININE (Investigations) | 1 | 0 | 0 | 0
BLOOD GLUCOSE FLUCTUATION (Investigations) | 1 | 0 | 0 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 0 | 1 | 0 | 0
BRONCHOSCOPY (Investigations) | 1 | 0 | 0 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0 | 0 | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 1 | 0 | 0 | 0
TROPONIN I INCREASED (Investigations) | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
DIABETIC FOOT (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 | 3 | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OBESITY (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 8 | 5 | 1 | 0
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 0
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 1
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 7 | 7 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 29 | 25 | 7 | 5
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 1
SPONDYLOARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 0
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 1 | 0
BENIGN DUODENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 2 | 0
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 0 | 1
BREAST CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
CARCINOID TUMOUR OF THE SMALL BOWEL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
CARDIAC MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
CHRONIC MYELOMONOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 3 | 1
EXTRANODAL MARGINAL ZONE B-CELL LYMPHOMA (MALT TYPE) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
INTRAVASCULAR PAPILLARY ENDOTHELIAL HYPERPLASIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
LANGERHANS' CELL GRANULOMATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
LENTIGO MALIGNA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LIP NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
LUNG CARCINOMA CELL TYPE UNSPECIFIED RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 1 | 4
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
MALIGNANT MELANOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
NEOPLASM PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
NON-SMALL CELL LUNG CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 10 | 0 | 0
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
SIGNET-RING CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 0
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 1
ANOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1 | 0 | 0
APHASIA (Nervous system disorders) | 0 | 1 | 0 | 0
ATAXIA (Nervous system disorders) | 1 | 1 | 0 | 0
BENIGN INTRACRANIAL HYPERTENSION (Nervous system disorders) | 0 | 0 | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 8 | 6 | 1 | 1
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 | 0 | 0 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0 | 0
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 0 | 2
DEMENTIA (Nervous system disorders) | 0 | 3 | 0 | 0
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 1 | 0 | 1 | 0
DEMYELINATION (Nervous system disorders) | 0 | 1 | 0 | 0
DIABETIC NEUROPATHY (Nervous system disorders) | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 5 | 4 | 0 | 3
ENCEPHALOPATHY (Nervous system disorders) | 1 | 1 | 0 | 0
FACIAL PALSY (Nervous system disorders) | 0 | 1 | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 2 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 1 | 2 | 0 | 2
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 | 0 | 0 | 1
INTRACRANIAL HYPOTENSION (Nervous system disorders) | 1 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 0 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1 | 0 | 1
MIGRAINE (Nervous system disorders) | 1 | 0 | 0 | 0
MYOCLONUS (Nervous system disorders) | 1 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 0 | 1 | 0
PERONEAL NERVE PALSY (Nervous system disorders) | 1 | 0 | 0 | 0
POST HERPETIC NEURALGIA (Nervous system disorders) | 1 | 0 | 0 | 0
POST-TRAUMATIC EPILEPSY (Nervous system disorders) | 0 | 1 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 2 | 0 | 0
RADICULOPATHY (Nervous system disorders) | 0 | 1 | 0 | 0
REVERSIBLE POSTERIOR LEUKOENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 2 | 0 | 0
SENSORY DISTURBANCE (Nervous system disorders) | 0 | 1 | 0 | 0
SPINAL CLAUDICATION (Nervous system disorders) | 1 | 0 | 0 | 0
SPINAL CORD DISORDER (Nervous system disorders) | 1 | 0 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 10 | 9 | 7 | 3
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 4 | 8 | 1 | 2
VASCULAR DEMENTIA (Nervous system disorders) | 0 | 0 | 0 | 1
VERTEBRAL ARTERY OCCLUSION (Nervous system disorders) | 1 | 0 | 0 | 0
PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
ALCOHOL WITHDRAWAL SYNDROME (Psychiatric disorders) | 1 | 0 | 0 | 0
ALCOHOLISM (Psychiatric disorders) | 1 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 1 | 1 | 0 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 1 | 1 | 1
CONVERSION DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0
DELIRIUM TREMENS (Psychiatric disorders) | 0 | 0 | 0 | 1
DELUSION (Psychiatric disorders) | 0 | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 2 | 2 | 0 | 0
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 0 | 1 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 1 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 2 | 0 | 2
PARANOIA (Psychiatric disorders) | 1 | 0 | 0 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0
SUICIDAL IDEATION (Psychiatric disorders) | 1 | 1 | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1 | 0 | 0
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0 | 0
BLADDER MASS (Renal and urinary disorders) | 0 | 1 | 0 | 0
BLADDER OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0 | 1
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 1 | 1 | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 4 | 0 | 0 | 0
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 0 | 1 | 0 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 2 | 0 | 1 | 0
HYDROURETER (Renal and urinary disorders) | 1 | 0 | 0 | 0
HYPERTONIC BLADDER (Renal and urinary disorders) | 0 | 1 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 3 | 4 | 0 | 0
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 4 | 1 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 1 | 1 | 0 | 0
RENAL CYST (Renal and urinary disorders) | 0 | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 2 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 12 | 7 | 2 | 2
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 | 1 | 1 | 1
URETERIC STENOSIS (Renal and urinary disorders) | 0 | 1 | 0 | 0
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 3 | 1 | 0
EPIDIDYMAL CYST (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
OVARIAN TORSION (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 14 | 11 | 6 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 2 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 0 | 0
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
DIABETIC ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 0 | 0 | 0 | 1
IMPLANTABLE DEFIBRILLATOR REPLACEMENT (Surgical and medical procedures) | 1 | 0 | 0 | 0
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 | 1 | 0 | 0
MITRAL VALVE REPLACEMENT (Surgical and medical procedures) | 0 | 0 | 0 | 1
ANEURYSM (Vascular disorders) | 1 | 0 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 5 | 1 | 1 | 0
AORTIC STENOSIS (Vascular disorders) | 4 | 2 | 0 | 2
AORTITIS (Vascular disorders) | 1 | 0 | 0 | 0
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1 | 0 | 0
ARTERIAL STENOSIS (Vascular disorders) | 0 | 0 | 1 | 0
ARTERIOSCLEROSIS (Vascular disorders) | 0 | 3 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 2 | 1 | 0
FEMORAL ARTERIAL STENOSIS (Vascular disorders) | 2 | 0 | 0 | 0
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 1 | 0 | 0
HAEMATOMA (Vascular disorders) | 2 | 1 | 2 | 1
HYPERTENSION (Vascular disorders) | 4 | 4 | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 3 | 1 | 0
HYPERTENSIVE EMERGENCY (Vascular disorders) | 1 | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 2 | 1 | 0 | 1
ILIAC ARTERY OCCLUSION (Vascular disorders) | 1 | 0 | 0 | 0
INTERMITTENT CLAUDICATION (Vascular disorders) | 7 | 1 | 0 | 0
ISCHAEMIA (Vascular disorders) | 0 | 1 | 0 | 0
MALIGNANT HYPERTENSION (Vascular disorders) | 2 | 1 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0
PELVIC VENOUS THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 5 | 2 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 3 | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 4 | 1 | 3
SUBCLAVIAN ARTERY STENOSIS (Vascular disorders) | 1 | 0 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0 | 0
THROMBOSIS (Vascular disorders) | 1 | 0 | 0 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 1 | 0 | 0
VASCULAR CALCIFICATION (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCRI DAPT - DES 30-month DAPT (N=0) | HCRI DAPT - DES 12-month DAPT (N=0) | HCRI DAPT - BMS 30-month DAPT (N=0) | HCRI DAPT - BMS 12-month DAPT (N=0)
AEs were not collected in the DAPT Trial (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — AEs that did not meet serious criteria were not routinely collected and reported by the investigators (only if they resulted in study discontinuation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No